CLINICAL TRIAL: NCT04776772
Title: Differential Health Effects on Inflammatory, Immunological and Stress Parameters in Professional Soccer Players and Sed-entary Individuals After Consuming a Synbiotic. A Triple Blind-ed, Randomized, Placebo-controlled Pilot Study
Brief Title: Health Parameters in Soccer Players and Sedentary Individuals After Consuming a Synbiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Murcia (Other)
Responsible Party: Principal Investigator, Carmen Daniela Quero Calero, Professor, principal investigator, Catholic University of Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CE031810
Record Dates: First submitted 2021-02-08; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Athlete; Sedentary Behavior
Keywords: anxiety; immunity; inflammation; prebiotic; probiotic; sedentarism; soccer; stress; synbiotic
MeSH Terms: conditions — Sedentary Behavior; Anxiety Disorders; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soccer player placebo (Placebo Comparator): Soccer player consuming placebo sticks filled with 300 mg excipient of maltodextrin
  Interventions: Dietary Supplement: Placebo
- Soccer player synbiotic (Experimental): Soccer players consuming a mixture of probiotic strains: Bifidobacterium lactis CBP-001010, Lactobacillus rhamno-sus CNCM I-4036, Bifidobacterium longum ES1 and fructooligosaccharides (200 mg) as a prebiotic
  Interventions: Dietary Supplement: Synbiotic complement
- Sedentary individuals placebo (Placebo Comparator): Sedentary individuals consuming placebo sticks filled with 300 mg excipient of maltodextrin
  Interventions: Dietary Supplement: Placebo
- Sedentary individuals synbiotic (Experimental): Sedentary individuals consuming a mixture of probiotic strains: Bifidobacterium lactis CBP-001010, Lactobacillus rhamno-sus CNCM I-4036, Bifidobacterium longum ES1 and fructooligosaccharides (200 mg) as a prebiotic
  Interventions: Dietary Supplement: Synbiotic complement

INTERVENTIONS:
Dietary Supplement: Synbiotic complement — On two separate days, the "baseline-tests" and "final-tests" were conducted. All participants performed a series of tests, before which they had to fast. The order and schedule (8 am) of the tests was the same for the "final-test" and the same materials and procedures were used. A period of 30 consecutive days elapsed between the base-line and final tests, during which the participants had to ingest their supplement (synbiotic).
  Arms: Sedentary individuals synbiotic; Soccer player synbiotic
Dietary Supplement: Placebo — On two separate days, the "baseline-tests" and "final-tests" were conducted. All participants performed a series of tests, before which they had to fast. The order and schedule (8 am) of the tests was the same for the "final-test" and the same materials and procedures were used. A period of 30 consecutive days elapsed between the base-line and final tests, during which the participants had to ingest their supplement (placebo).
  Arms: Sedentary individuals placebo; Soccer player placebo

SUMMARY:
The main objective of this research was to carry out an experimental study, triple blind, on the possible immunophysiological effects of a nutritional supplement (Synbiotic, Gasteel Plus®, Heel España S.A.U.), containing a mixture of probiotic strains, such as Bifidobacterium lactis CBP-001010, Lactobacillus rhamnosus CNCM I-4036, Bifidobacterium longum ES1, as well as prebi-otic fructooligosaccharides, in both professional athletes and sedentary people. The effects on some inflammatory/immune (IL-1β, IL-10, and immunoglobulin A) and stress (epinephrine, nore-pinephrine, dopamine, serotonin, CRH, ACTH, and cortisol) biomarkers were evaluated, determined by flow cytometer and ELISA. The effects on metabolic profile and physical activity, as well as on various parameters that could affect physical and mental health, were also evaluated via the use of accelerometry and validated questionnaires.

DETAILED DESCRIPTION:
This investigation was a triple blinded, randomized, placebo-controlled pilot study designed to identify the possible differing effects of the synbiotic Gasteel Plus® supplementation.

The participants were professional soccer players of the Second Division B of the Spanish League and sedentary students of the same sex and age range. Both study groups were randomly divided into two groups: a control group administered with placebo, and an experimental group administered with the synbiotic. Each participant was evaluated at baseline, as well as after the intervention which lasted one month. Only in the athletes group did the synbiotic intervention clearly improve objective physical activ-ity and sleep quality, as well as perceived general health, stress, and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals: students with low levels of physical activity (≤ 150 minutes/week),
* Athletes: semi professional soccer players

Exclusion Criteria:

* Participants were prohibited from consuming probiotics, prebiotics or fermented products (yogurt or other foods)
* Presenting injury or illness

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Objective determination of levels of physical activity, sedentary lifestyle and sleep quality: accelerometry | During 7 days before the ingestion of the synbiotic or placebo
  Participants wore the accelerometer held with an elastic band on the non-dominant wrist for 7 consecutive days and without interruption, except for those times of the day in which the correct operation of the device could be compromised (showers or any activity related to wa-ter). Subsequently, the files generated by the accelerometer were analyzed through a specific software called Actilife 6 (Actigraph, Pensacola, USA).
Objective determination of levels of physical activity, sedentary lifestyle and sleep quality: accelerometry | During 7 days after the ingestion of the synbiotic or placebo
  Participants wore the accelerometer held with an elastic band on the non-dominant wrist for 7 consecutive days and without interruption, except for those times of the day in which the correct operation of the device could be compromised (showers or any activity related to wa-ter). Subsequently, the files generated by the accelerometer were analyzed through a specific software called Actilife 6 (Actigraph, Pensacola, USA).
Questionnarie about general health. | One day before the ingestion of the synbiotic or placebo
  SF-36 Questionnaire: Scale from 0 to 100. Higher scores mean a better outcome.
Questionnarie about general health. | One day after the ingestion of the synbiotic or placebo
  SF-36 Questionnaire: Scale from 0 to 100. Higher scores mean a better outcome.
Questionnarie about anxiety levels (moment) | One day before the ingestion of the synbiotic or placebo
  The State Anxiety Inventory (STAI): Scale from 0 to 60. Higher scores mean a worse outcome.
Questionnarie about anxiety levels (moment) | One day after the ingestion of the synbiotic or placebo
  The State Anxiety Inventory (STAI): Scale from 0 to 60. Higher scores mean a worse outcome.
Questionnarie about anxiety levels (personality) | One day before the ingestion of the synbiotic or placebo
  The Trait Anxiety Inventory (STAI): Scale from 0 to 60. Higher scores mean a worse outcome.
Questionnarie about anxiety levels (personality) | One day after the ingestion of the synbiotic or placebo
  The Trait Anxiety Inventory (STAI): Scale from 0 to 60. Higher scores mean a worse outcome.
Questionnarie about sleep quality | One day before the ingestion of the synbiotic or placebo
  Healthy Lifestyle and Personal Control Questionnaire: Scale from -1 to 10. Higher scores mean a better outcome.
Questionnarie about sleep quality | One day after the ingestion of the synbiotic or placebo
  Healthy Lifestyle and Personal Control Questionnaire: Scale from -1 to 10. Higher scores mean a better outcome.
Questionnarie about perceived stress | One day before the ingestion of the synbiotic or placebo
  The Perceived Stress Scale: Scale from 0 to 56. Higher scores mean a worse outcome.
Questionnarie about perceived stress | One day after the ingestion of the synbiotic or placebo
  The Perceived Stress Scale: Scale from 0 to 56. Higher scores mean a worse outcome.
Questionnarie about perceived fatigue | One day before the ingestion of the synbiotic or placebo
  Brief Fatigue Inventory: Scale from 0 to 40. Higher scores mean a worse outcome.
Questionnarie about perceived fatigue | One day after the ingestion of the synbiotic or placebo
  Brief Fatigue Inventory: Scale from 0 to 40. Higher scores mean a worse outcome.
Questionnarie about perceived depression | One day before the ingestion of the synbiotic or placebo
  Beck´s Depression Inventory: Scale from 0 to 63. Higher scores mean a worse outcome.
Questionnarie about perceived depression | One day after the ingestion of the synbiotic or placebo
  Beck´s Depression Inventory: Scale from 0 to 63. Higher scores mean a worse outcome.
Determination of the pro-inflammatory cytokine IL-1β (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Using the LuminexTM 200 System instrument (Luminex Corporation, Texas, USA) using the ProcartaPlex TM Multiplex Immunoassay for analysis.
  Measured in pg/ml.
Determination of the pro-inflammatory cytokine IL-1β (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Using the LuminexTM 200 System instrument (Luminex Corporation, Texas, USA) using the ProcartaPlex TM Multiplex Immunoassay for analysis.
  Measured in pg/ml.
Determination of the anti-inflammatory cytokine IL-10 (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Using the LuminexTM 200 System instrument (Luminex Corporation, Texas, USA) using the ProcartaPlex TM Multiplex Immunoassay for analysis.
  Measured in pg/ml.
Determination of the anti-inflammatory cytokine IL-10 (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Using the LuminexTM 200 System instrument (Luminex Corporation, Texas, USA) using the ProcartaPlex TM Multiplex Immunoassay for analysis.
  Measured in pg/ml.
Determination of the stress hormones Cortisol (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The DetectX Cortisol Immunoassay Kit.
  Measured in µg/dl.
Determination of the stress hormones Cortisol (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The DetectX Cortisol Immunoassay Kit.
  Measured in µg/dl.
Determination of the adrenocorticotropic hormone (ACTH) (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Human ACTH (Adrenocorticotropic Hormone) ELISA Kit (Elabscience, USA).
  Measured in pg/ml.
Determination of the adrenocorticotropic hormone (ACTH) (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Human ACTH (Adrenocorticotropic Hormone) ELISA Kit (Elabscience, USA).
  Measured in pg/ml.
Determination of the corticotropin-releasing hormone (CRH) (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Human Corticotropin Releasing Hormone (CRH) RD-CRH-Hu (Kelowna, BC, V1W 4V3, Canada) Measured in pg/ml.
Determination of the corticotropin-releasing hormone (CRH) (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Human Corticotropin Releasing Hormone (CRH) RD-CRH-Hu (Kelowna, BC, V1W 4V3, Canada) Measured in pg/ml.
Determination of the stress hormones serotonin (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General 5-Hydroxytryptamine (5-HT) RD-5-HT-Ge.
  Measured in ng/ml.
Determination of the stress hormones serotonin (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General 5-Hydroxytryptamine (5-HT) RD-5-HT-Ge.
  Measured in ng/ml.
Determination of the catecholamine dopamine (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Dopamine Research Immunoassay Measured in ng/ml.
Determination of the catecholamine dopamine (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The Dopamine Research Immunoassay Measured in ng/ml.
Determination of the catecholamine epinephrine (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General Epinephrine (EPI) RD-EPI-Ge-96T.
  Measured in pg/ml.
Determination of the catecholamine epinephrine (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General Epinephrine (EPI) RD-EPI-Ge-96T.
  Measured in pg/ml.
Determination of the catecholamine norepinephrine (Blood sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General Noradrenaline (NE) RD-NE-Ge-96T.
  Measured in pg/ml.
Determination of the catecholamine norepinephrine (Blood sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by competitive inhibition enzyme immunoassays (ELISA), using The General Noradrenaline (NE) RD-NE-Ge-96T.
  Measured in pg/ml.
Determination of the immunoglobulin A (Saliva sampling) | One day before the ingestion of the synbiotic or placebo
  Analyzed by indirect enzyme immunoassay kit through the Salivary Secretory IgA Kit (Salimetrics LLC, USA). The procedures followed the instructions of the manufacturers, and the findings were measured using an ELISA auto analyzer to quantify color intensity (Sunrise, Tecan, Männendorf, Switzerland).
  Measured in µg/ml
Determination of the immunoglobulin A (Saliva sampling) | One day after the ingestion of the synbiotic or placebo
  Analyzed by indirect enzyme immunoassay kit through the Salivary Secretory IgA Kit (Salimetrics LLC, USA). The procedures followed the instructions of the manufacturers, and the findings were measured using an ELISA auto analyzer to quantify color intensity (Sunrise, Tecan, Männendorf, Switzerland).
  Measured in µg/ml
Determination of glucose levels (metabolic profile) | One day before the ingestion of the synbiotic or placebo
  The determinations for obtaining the glycemic profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl
Determination of glucose levels (metabolic profile) | One day after the ingestion of the synbiotic or placebo
  The determinations for obtaining the glycemic profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl
Determination of total cholesterol levels (metabolic profile) | One day before the ingestion of the synbiotic or placebo
  The determinations for obtaining the lipid profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl
Determination of total cholesterol levels (metabolic profile) | One day after the ingestion of the synbiotic or placebo
  The determinations for obtaining the lipid profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl
Determination of the triglycerides levels (metabolic profile) | One day before the ingestion of the synbiotic or placebo
  The determinations for obtaining the lipid profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl
Determination of the triglycerides levels (metabolic profile) | One day after the ingestion of the synbiotic or placebo
  The determinations for obtaining the lipid profile were carried out through standard techniques with the automatic analyzer of clinical chemistry BA 400 (BioSystems) in the SYNLAB laboratories (Diagnosticos Globales S.A.U., Badajoz, Spain).
  Measured in mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Quero, PhD, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The raw data supporting the conclusions of this intervention will be made available by the investigators, without undue reservation, to any qualified researcher
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be always available upon reasonable request
Access Criteria: The data that support the findings of this study are available via email from the corresponding author upon reasonable request.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04776772/Prot_SAP_ICF_000.pdf